CLINICAL TRIAL: NCT04767633
Title: Randomized Controlled Trial Comparing Split-versus Standard-dose Sodium Pico Sulfate Plus Magnesium Citrate for Bowel Cleansing Before Colonoscopy in Children
Brief Title: Picoprep Split-dose Before Colonoscopy in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera "Sant'Andrea" (Other)
Responsible Party: Principal Investigator, Dr. Enrico Felici, Head of Pediatric Unit, Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PICOPREP-SPLIT v.1 02/09/2020
Record Dates: First submitted 2020-12-29; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Sodium Picosulfate Overdose; Magnesium Sulfate Overdose; Children, Only; Bowel Disease
MeSH Terms: conditions — Intestinal Diseases | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (PMC standard-dose) (Active Comparator): Group A (PMC standard-dose): patients will receive two oral doses of sodium picosulphate plus magnesium oxide and citric acid (Picoprep), each diluted in 150 ml of water, at 17:00 and 4 hours later in the evening prior to the colonoscopy (¼ sachet for children < 6 years, ½ sachet for children 6-12 years, and one sachet for children >12 years). Intake of at least 40-50 ml/kg (maximum 2 L) of clear fluids (cold tea, gatorade etc..) will be recommended after each dose. The age-adjusted dosage is dictated by the instructions of the manufacturing company. No solid food intake will be allowed during the 24 hours prior to the examination according to the instructions of the manufacturing company.
  Interventions: Drug: split dose vs standard dose of sodium pico sulfate plus magnesium sulfate in children for bowel cleansing
- Group B (PMC split-dose) (Active Comparator): Group B (PMC split-dose): patients will receive the first oral doses of PMC diluted in 150 ml of water (Picoprep; Ferring Italia, Milan, Italy) at 19:00 of the day before colonoscopy and the second one at 06:00 hours on the morning of the day of colonoscopy (¼ sachet for children < 6 years, ½ sachet for children 6-12 years, and one sachet for children >12 years). Intake of at least 40-50 ml/kg (maximum 2 L) of clear fluids (cold tea, gatorade etc..) will be recommended after each dose. The age-adjusted dosage is dictated by the instructions of the manufacturing company. No solid food intake will be allowed during the 24 hours prior to the examination according to the instructions of the manufacturing company.
  Interventions: Drug: split dose vs standard dose of sodium pico sulfate plus magnesium sulfate in children for bowel cleansing

INTERVENTIONS:
Drug: split dose vs standard dose of sodium pico sulfate plus magnesium sulfate in children for bowel cleansing — The preparations will be dispensed by a nurse who carefully explained how the products should be taken, emphasising the importance of complete intake of the solution to ensure a safe and effective procedure. Moreover, each patient will be provided with dietary instructions: low residue diet for 3 days before colonoscopy. During and after bowel preparation, solid food will not be allowed. Clear liquid could be taken until 2 hours before the procedure. All colonoscopy will be performed between 11:00 and 15:00 by two endoscopists.

SUMMARY:
Before having a colonoscopy, it is necessary to clean the intestine well in order to have a complete view of the intestinal mucosa. Preparations consisting of osmotic agents are used to clean the intestines, which are sometimes difficult to drink. In this study we want to evaluate whether the preparation, based on sodium picosulfate plus magnesium citrate (PMC), is easier for the patient to take all day before the exam or half the day before and half the same morning of procedure and which method of intake allows the doctor to better conduct the examination.

The primary objective of this study will be to compare the efficacy, tolerability and acceptability of two dosage regimens of sodium picosulfate plus magnesium citrate (PMC). Effectiveness means which of the two methods of taking the preparation works best for cleaning the intestine, with tolerability if one of the two methods is easier for the patient and with acceptability if one of the two methods is easier than the other.

DETAILED DESCRIPTION:
The primary aim of this investigator-blinded, randomized, controlled trial (RCT) will be to compare the efficacy, tolerability and acceptability of two PMC dosing regimen (standard regimen vs split-dose regimen).

The secondary aims are the following:

* evaluation of adverse events;
* assessment of symptoms associated to colonic lavage solutions;
* monitoring the ease of taking the preparation;
* identification of patients' willingness to repeat the procedure;
* evaluation of the amount of preparation voluntarily taken by patients.

Endpoints

Primary end-points will be the overall colon cleansing defined as the rate of "successful" cleansing (excellent and good scores in the BBPS, i.e. ≥ 6 points) of the two preparation regimen.

Secondary end-points will include: 1) the rate of adverse events, 2) the rate of specific

symptoms associated to colonic lavage solutions, 3) the rate of children who declared that the intake of the solution was easy, 4) the rate of children who declared that they would be willing to repeat the same preparation regimen if needed, 5) the rate of children taking an amount of solution ≥ 75%.

PATIENTS AND METHODS

Study design

This will be a multicenter, randomized, non-pharmacological, observer-blind, parallel group study conducted in Italy.

The study is considered non-pharmacological because we'll use the standard dose administered with two different timing (assumption of the whole preparation on the day prior to investigative procedure vs assumption of the first half of oral doses the day before colonoscopy and the second one on the morning of the day of colonoscopy).

The patients enrolled will be randomized in one of the two arms that provide the following treatment:

Group A: they will receive PCM standard-dose which provides for the assumption of whole dose of preparation on the day prior to investigative procedure; Group B: they will receive PCM split-dose administered the previous day and in the morning of the day of colonoscopy.

Study period

The total duration of this study is expected to be 18 months from the approval of the ethical committee assuming an expected enrollment duration of 16 months.

Adverse events will be assessed on the day of colonoscopy by direct questioning and by telephone interview 48-96 hours after colonoscopy.

Participants

Eligible participants will be all consecutive children aged 2-18 years undergoing elective colonoscopy in the involved institutions with informed consent signed by the parent/ guardian. Exclusion criteria are: 1) requirement for urgent colonoscopy, 2) bowel obstruction, 3) known or suspected hypersensitivity to the active or other ingredients, 4) clinically significant electrolyte imbalance, 5) prior intestinal resection, 6) known metabolic, renal and cardiac disease.

Written assent from young patients and informed consent from the legal guardian and patients over fourteen years will be obtained

Interventions

Group A (PMC standard-dose): patients will receive two oral doses of sodium picosulphate plus magnesium oxide and citric acid (Picoprep), each diluted in 150 ml of water, at 17:00 and 4 hours later in the evening prior to the colonoscopy (¼ sachet for children < 6 years, ½ sachet for children 6-12 years, and one sachet for children >12 years). Intake of at least 40-50 ml/kg (maximum 2 L) of clear fluids (cold tea, gatorade etc..) will be recommended after each dose. The age-adjusted dosage is dictated by the instructions of the manufacturing company. No solid food intake will be allowed during the 24 hours prior to the examination according to the instructions of the manufacturing company.

Group B (PMC split-dose): patients will receive the first oral doses of PMC diluted in 150 ml of water (Picoprep; Ferring Italia, Milan, Italy) at 19:00 of the day before colonoscopy and the second one at 06:00 hours on the morning of the day of colonoscopy (¼ sachet for

children < 6 years, ½ sachet for children 6-12 years, and one sachet for children >12 years). Intake of at least 40-50 ml/kg (maximum 2 L) of clear fluids (cold tea, gatorade etc..) will be recommended after each dose. The age-adjusted dosage is dictated by the instructions of the manufacturing company. No solid food intake will be allowed during the 24 hours prior to the examination according to the instructions of the manufacturing company.

In both groups a nasogastric tube will be inserted if the child failed to drink the prescribed amount of cleanout preparation within the first hour.

The preparations will be dispensed by a nurse who carefully explained how the products should be taken, emphasising the importance of complete intake of the solution to ensure a safe and effective procedure. Moreover, each patient will be provided with dietary instructions: low residue diet for 3 days before colonoscopy. During and after bowel preparation, solid food will not be allowed. Clear liquid could be taken until 2 hours before the procedure. All colonoscopy will be performed between 11:00 and 15:00 by two endoscopists.

Evaluation of bowel preparations

Efficacy. Preparation efficacy will be evaluated by the blinded endoscopist according to the Boston Bowel Preparation scale (BBPS) (14) consisting of four-point scoring system applied to each of the three broad regions of the colon: right colon, transverse colon, and left colon In addition, overall cleansing of the colon will be scored by summing up the scores of each segment. For the study, the total score ranging from 0 to 9 will be divided into four different classes: excellent cleansing (total score 8-9), good cleansing (total score 6-7), poor cleansing (total score 4-5) and inadequate cleansing (total score 0-3). For the primary efficacy variable, excellent and good cleansing will be considered as "successful" and poor or inadequate as "failure".

According with a normal clinical practice, all examinations will be performed with a pediatric colonoscope under general anesthesia.

Safety. Vital signs, complete physical examination and routine blood tests will be performed at the time of patient enrolment and on the day of colonoscopy and included liver and kidney function test, potassium, magnesium, sodium, chlorides and calcium. Adverse events will be assessed on the day of colonoscopy by direct questioning and by telephone interview 48-96 hours after colonoscopy. All new symptoms will be considered to be treatment related and have been included in the analysis. Any symptom that manifested following the treatment (except those expected and included in the evaluation of GI- tolerability) and exacerbations of preexisting symptoms will be assumed to be related to the bowel preparation regimen.

Tolerability, acceptability and compliance. On the morning of colonoscopy, immediately before the procedure, a nurse questioned each patient about his/her experience by using a standardized questionnaire (see below). Patients will be inquired about tolerability, need for nasogastric tube placement, acceptability and compliance. The endoscopist will not be allowed to take part in the questioning or to supervise the clinical interview before colonoscopy.

Tolerability assessment will be based on the recording of occurrence and severity of GI symptoms such as nausea, bloating, abdominal, pain/cramps and anal discomfort. A 5-point scale (1 = severely distressing, 2 = distressing, 3 = bothersome, 4 = mild and 5 = none), will be used to score the tolerability (10). The need for nasogastric tube insertion will also be assessed.

The easiness of taking or swallowing the solution will be graded according to the following scale: very severe distress = 4, severe distress = 3, moderate distress = 2, mild distress = 1, no distress = 0.

Willingness to repeat the same type of bowel preparation if necessary will also be evaluated. Compliance will be scored on a 3-point scale according to the percentage of drunken solution (excellent: intake of the whole solution; good: intake of at least 75% of the solution; poor: intake of < 75%).

Randomization and blinding

A randomised computer-generated list in blocks of six will be prepared by a biostatistician and eligible children were allocated to receive one of the two bowel preparations, stratified by three age groups; 2-7 years, 8-13 years and 14-18 years. A clinic nurse will assign treatment regimen only after written consent will be obtained by one of the investigators. The cleanout regimen will be dispensed directly to the family.

The study will be observer blind: the endoscopists will not be allowed to perform any activities associated with study preparation prior and after colonoscopy and will avoid any discussion with the patients and the staff, which could disclose the type of bowel preparation.

Statistical Analysis

Based on results from previous studies on bowel preparation with PMC on adults patients, a success rate of about 75 % was assumed (15) difference in efficacy of 10% (80% in split-dose vs. 70% in single dose) between the two groups, with power of study 80%, alpha error 0.05 and confidence interval 95% calculated sample size will be 290 patients in each arm.

For univariate analysis, comparisons between groups will be performed using the Student's t test, the chi-squared test, or Fisher's exact test, as appropriate. The Mann - Whitney test will be used to compare non-paired, nonparametric variables. Multivariate analysis will be used for the primary outcome variables, in a logistic step- wise regression model. The statistical analysis will be performed using absolute and relative frequency tables and contingency

tables. The statistical significance will be set at p < 0.05. The analysis will be conducted using SPSS, release 23.0 version.

ELIGIBILITY:
Inclusion Criteria:

• children aged 2-18 years undergoing elective colonoscopy

Exclusion Criteria:

* requirement for urgent colonoscopy
* bowel obstruction,
* known or suspected hypersensitivity to the active or other ingredients
* clinically significant electrolyte imbalance
* prior intestinal resection
* known metabolic, renal and cardiac disease.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 590 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-04-16 (Estimated); Study Completion 2022-07-16 (Estimated)

PRIMARY OUTCOMES:
Best Colonic Cleansing in 590 pediatric patient underwent colonoscopy | 18 months
  Primary outcome will be the overall colon cleansing defined as the rate of successful cleansing (excellent and good scores in the BBPS, i.e. ≥ 6 points) of the two preparation regimen.

SECONDARY OUTCOMES:
the rate of adverse events | 18 months
  Percentage of adverse events between two preparation regimen
the rate of specific symptoms associated to colonic lavage solutions | 18 months
  percentage of symptoms associated to bowel preparation
the rate of children who declared that they would be willing to repeat the same preparation regimen if needed | 18 months
  percentage of children well tollerate the praparation taken
the rate of children who declared that the intake of the solution was easy | 18 months
  percentage of children not discomfort to drink solution
the rate of children taking an amount of solution ≥ 75% | 18 months
  Percentage of patient take sufficient dose of bowel preparation

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Felici, DR, Principal Investigator — Azienda Ospedaliera SS. Antonio e Biagio e C. Arrigo - Alessandria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ASGE Standards of Practice Committee; Lightdale JR, Acosta R, Shergill AK, Chandrasekhara V, Chathadi K, Early D, Evans JA, Fanelli RD, Fisher DA, Fonkalsrud L, Hwang JH, Kashab M, Muthusamy VR, Pasha S, Saltzman JR, Cash BD; American Society for Gastrointestinal Endoscopy. Modifications in endoscopic practice for pediatric patients. Gastrointest Endosc. 2014 May;79(5):699-710. doi: 10.1016/j.gie.2013.08.014. Epub 2014 Mar 1. PMID 24593951
- [Background] Froehlich F, Wietlisbach V, Gonvers JJ, Burnand B, Vader JP. Impact of colonic cleansing on quality and diagnostic yield of colonoscopy: the European Panel of Appropriateness of Gastrointestinal Endoscopy European multicenter study. Gastrointest Endosc. 2005 Mar;61(3):378-84. doi: 10.1016/s0016-5107(04)02776-2. PMID 15758907
- [Background] Belsey J, Epstein O, Heresbach D. Systematic review: oral bowel preparation for colonoscopy. Aliment Pharmacol Ther. 2007 Feb 15;25(4):373-84. doi: 10.1111/j.1365-2036.2006.03212.x. PMID 17269992
- [Background] Barkun A, Chiba N, Enns R, Marcon M, Natsheh S, Pham C, Sadowski D, Vanner S. Commonly used preparations for colonoscopy: efficacy, tolerability, and safety--a Canadian Association of Gastroenterology position paper. Can J Gastroenterol. 2006 Nov;20(11):699-710. doi: 10.1155/2006/915368. PMID 17111052
- [Background] Dahshan A, Lin CH, Peters J, Thomas R, Tolia V. A randomized, prospective study to evaluate the efficacy and acceptance of three bowel preparations for colonoscopy in children. Am J Gastroenterol. 1999 Dec;94(12):3497-501. doi: 10.1111/j.1572-0241.1999.01613.x. PMID 10606310
- [Background] Hunter A, Mamula P. Bowel preparation for pediatric colonoscopy procedures. J Pediatr Gastroenterol Nutr. 2010 Sep;51(3):254-61. doi: 10.1097/MPG.0b013e3181eb6a1c. PMID 20683200
- [Background] Pall H, Zacur GM, Kramer RE, Lirio RA, Manfredi M, Shah M, Stephen TC, Tucker N, Gibbons TE, Sahn B, McOmber M, Friedlander J, Quiros JA, Fishman DS, Mamula P. Bowel preparation for pediatric colonoscopy: report of the NASPGHAN endoscopy and procedures committee. J Pediatr Gastroenterol Nutr. 2014 Sep;59(3):409-16. doi: 10.1097/MPG.0000000000000447. PMID 24897169
- [Background] Hassan C, East J, Radaelli F, Spada C, Benamouzig R, Bisschops R, Bretthauer M, Dekker E, Dinis-Ribeiro M, Ferlitsch M, Fuccio L, Awadie H, Gralnek I, Jover R, Kaminski MF, Pellise M, Triantafyllou K, Vanella G, Mangas-Sanjuan C, Frazzoni L, Van Hooft JE, Dumonceau JM. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2019. Endoscopy. 2019 Aug;51(8):775-794. doi: 10.1055/a-0959-0505. Epub 2019 Jul 11. PMID 31295746
- [Background] Tripathi PR, Poddar U, Yachha SK, Sarma MS, Srivastava A. Efficacy of Single- Versus Split-dose Polyethylene Glycol for Colonic Preparation in Children: A Randomized Control Study. J Pediatr Gastroenterol Nutr. 2020 Jan;70(1):e1-e6. doi: 10.1097/MPG.0000000000002511. PMID 31567887
- [Background] Sriphongphankul H, Tanpowpong P, Lertudomphonwanit C, Treepongkaruna S. Split dose versus full single-dose regimen of polyethylene glycol for bowel preparation in pediatric colonoscopy: a pilot study of randomized controlled trial. Eur J Gastroenterol Hepatol. 2019 Nov;31(11):1382-1386. doi: 10.1097/MEG.0000000000001562. PMID 31567637
- [Background] Martel M, Barkun AN, Menard C, Restellini S, Kherad O, Vanasse A. Split-Dose Preparations Are Superior to Day-Before Bowel Cleansing Regimens: A Meta-analysis. Gastroenterology. 2015 Jul;149(1):79-88. doi: 10.1053/j.gastro.2015.04.004. Epub 2015 Apr 8. PMID 25863216
- [Background] Di Nardo G, Aloi M, Cucchiara S, Spada C, Hassan C, Civitelli F, Nuti F, Ziparo C, Pession A, Lima M, La Torre G, Oliva S. Bowel preparations for colonoscopy: an RCT. Pediatrics. 2014 Aug;134(2):249-56. doi: 10.1542/peds.2014-0131. Epub 2014 Jul 7. PMID 25002661
- [Background] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102
- [Background] Manes G, Repici A, Hassan C; MAGIC-P study group. Randomized controlled trial comparing efficacy and acceptability of split- and standard-dose sodium picosulfate plus magnesium citrate for bowel cleansing prior to colonoscopy. Endoscopy. 2014 Aug;46(8):662-9. doi: 10.1055/s-0034-1365800. Epub 2014 Jul 14. PMID 25019969